CLINICAL TRIAL: NCT02002052
Title: Functional Lung Avoidance for Individualized Radiotherapy (FLAIR): A Randomized, Double-Blind Clinical Trial
Acronym: FLAIR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWO-FLAIR
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer, radiotherapy, chemotherapy, pneumonitis, functional lung avoidance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Arm (Active Comparator): Standard platinum-based chemoradiotherapy, total radiation dose 60 Gy in 30 fractions
  Interventions: Drug: Concurrent platinum-based chemotherapy; Radiation: Standard Radiotherapy, 60 Gy in 30 fractions.
- Experimental Arm (Experimental): Functional-lung avoidance radiotherapy, total dose 60 Gy in 30 fractions, with concurrent platinum-based chemotherapy
  Interventions: Drug: Concurrent platinum-based chemotherapy; Radiation: Functional Lung Avoidance Radiotherapy, 60 Gy in 30 fractions

INTERVENTIONS:
Drug: Concurrent platinum-based chemotherapy — Platinum-based concurrent chemotherapy in both arms
Radiation: Standard Radiotherapy, 60 Gy in 30 fractions.
  Arms: Standard Arm
Radiation: Functional Lung Avoidance Radiotherapy, 60 Gy in 30 fractions
  Arms: Experimental Arm

SUMMARY:
Concurrent chemoradiotherapy is the standard treatment for locally advanced, unresectable non-small cell lung cancer, but carries a risk of radiation pneumonitis of approximately 30%, and is associated with a decline in pulmonary quality of life.

Standard radiation planning aims to optimize dose to the anatomic lung volume, without consideration of the differences in regional lung function. Functional lung avoidance radiotherapy aims to reduce radiotherapy dose to regions of functioning lung, instead depositing dose in areas of lung that are not well-ventilated. Functional lung regions are determined using noble-gas MRI and co-registered to the radiotherapy planning CT scans. Functional lung avoidance radiotherapy has been demonstrated to be feasible, and this trial aims to compare outcomes between standard radiotherapy (with concurrent chemotherapy) vs. functional lung avoidance radiotherapy (with concurrent chemotherapy).

DETAILED DESCRIPTION:
All consenting patients will undergo hyperpolarized noble gas MRI using 3-He for definition of functional lung volumes. Two radiotherapy treatment plans will be generated prior to randomization: one standard plan using anatomical lung avoidance, and one functional lung avoidance plan. After approval of both plans, patients will be randomized, and both patients and physicians will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed non-small cell lung carcinoma
* Locally advanced Stage IIIA or IIIB lung carcinoma according to AJCC 7th edition
* History of at least 10-pack-years of smoking
* Not undergoing surgical resection
* Assessment by medical oncologist and radiation oncologist, with adequate bone marrow, hepatic and renal function for administration of platinum-based chemotherapy

Exclusion Criteria:

* Contraindications to MRI
* Serious medical comorbidities (such as unstable angina, sepsis) or other contraindications to radiotherapy or chemotherapy
* Prior history of lung cancer within 5 years
* Prior thoracic radiation at any time
* Metastatic disease. Patients who present with oligometastatic disease where all metastases have been ablated (with surgery or radiotherapy) are candidates if they are receiving chemoradiotherapy to the thoracic disease with curative intent.
* Inability to attend full course of radiotherapy or follow-up visits
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary quality of life 3-months post-treatment. | 3-months post-treatment
  Measured using the Functional-Assessment of Cancer Therapy-Lung Cancer Subscale (FACT-LCS)

SECONDARY OUTCOMES:
Quality of life at other time points | up to 1 year
  Measured using the FACT-LCS, FACT-TOI, and FACT-L
Toxicity | up to 1 yr
  CTC-AE version 4
Overall Survival | 5-years
  Defined as time from randomization to death from any cause
Progression Free Survival | Up to 5 years
  Time from randomization to disease progression at any site or death
Quality-adjusted survival | Up to 5 years
  Based on utilities from EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Brian Yaremko, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Hoover DA, Capaldi DP, Sheikh K, Palma DA, Rodrigues GB, Dar AR, Yu E, Dingle B, Landis M, Kocha W, Sanatani M, Vincent M, Younus J, Kuruvilla S, Gaede S, Parraga G, Yaremko BP. Functional lung avoidance for individualized radiotherapy (FLAIR): study protocol for a randomized, double-blind clinical trial. BMC Cancer. 2014 Dec 11;14:934. doi: 10.1186/1471-2407-14-934. PMID 25496482